CLINICAL TRIAL: NCT01175785
Title: Infusion of Off-the-Shelf Ex Vivo Expanded Cryopreserved Cord Blood Progenitor Cells to Augment Single or Double Myeloablative Cord Blood Transplantation in Patients With Hematologic Malignancies
Brief Title: Infusion of Off-the-Shelf Expanded Cord Blood Cells to Augment Cord Blood Transplant in Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nohla Therapeutics, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2378.00; NCI-2010-01426 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2378; 2378.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); RC2HL101844 (NIH)
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Chronic Myelogenous Leukemia; Childhood Myelodysplastic Syndromes; Chronic Phase Chronic Myelogenous Leukemia; de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Refractory Anemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Excess Blasts in Transformation; Relapsing Chronic Myelogenous Leukemia; Secondary Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic-Phase; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts | interventions — Cord Blood Stem Cell Transplantation; Transplantation; fludarabine phosphate; Cyclophosphamide; Whole-Body Irradiation; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemo, radiation, transplant, GVHD prophylaxis) (Experimental): Patients receive fludarabine phosphate IV over 1 hour on days -8 to -6 and cyclophosphamide IV on days -7 and -6. Patients undergo TBI twice daily on days -4 to -1. Patients undergo unmanipulated single- or double-unit umbilical cord blood transplantation on day 0 and receive ex vivo-expanded cord blood progenitor cells IV over 4 hours following the last unmanipulated cord blood infusion. Patients initially receive CSP IV over 1 hour beginning on day -3. CSP may be given PO when the patient can tolerate oral medications and has a normal gastrointestinal transit time. CSP is given until day 100, and may taper on day 101 if there is no graft versus host disease. Patients also receive MMF IV every 8 hours on days 0 to 7 and then may receive MMF PO beginning day 8 to 30. MMF is continued for a minimum of 30 days or until 7 days after blood counts recover whichever is later. If there is no evidence of acute GVHD and donor CD3 engraftment is at least 50% from one donor MMF may be tapered.
  Interventions: Procedure: umbilical cord blood transplantation; Drug: fludarabine phosphate; Drug: cyclophosphamide; Biological: ex vivo-expanded cord blood progenitor cell infusion; Radiation: total-body irradiation; Drug: cyclosporine; Drug: mycophenolate mofetil; Other: laboratory biomarker analysis

INTERVENTIONS:
Procedure: umbilical cord blood transplantation — Undergo unmanipulated umbilical cord blood transplant
  Other Names: cord blood transplantation; transplantation, umbilical cord blood; UCB transplantation
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: ex vivo-expanded cord blood progenitor cell infusion — Undergo ex-vivo expanded cryopreserved cord blood progenitor cells
  Other Names: Dilanubicel; NLA101
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Drug: cyclosporine — Given IV
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: mycophenolate mofetil — Given IV and PO
  Other Names: Cellcept; MMF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying the safety and potential efficacy of infusing non-human leukocyte antigen matched ex vivo expanded cord blood progenitors with one or two unmanipulated umbilical cord blood units for transplantation following conditioning with fludarabine phosphate, cyclophosphamide and total body irradiation, and immunosuppression with cyclosporine and mycophenolate mofetil for patients with hematologic malignancies. Chemotherapy, such as fludarabine phosphate and cyclophosphamide, and total-body irradiation given before an umbilical cord blood transplant stops the growth of leukemia cells and works to prevent the patient's immune system from rejecting the donor's stem cells. The healthy stem cells from the donor's umbilical cord blood help the patient's bone marrow make new red blood cells, white blood cells, and platelets. It may take several weeks for these new blood cells to grow. During that period of time, patients are at increased risk for bleeding and infection. Faster recovery of white blood cells may decrease the number and severity of infections. Studies have shown that counts recover more quickly when more cord blood cells are given with the transplant. We have developed a way of growing or "expanding" the number of cord blood cells in the lab so that there are more cells available for transplant. We are doing this study to find out whether or not giving these expanded cells along with one or two unexpanded cord blood units is safe and if use of expanded cells can decrease the time it takes for white blood cells to recover after transplant. We will study the time it takes for blood counts to recover, which of the two or three cord blood units makes up the patient's new blood system, and how quickly immune system cells return.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the safety and toxicity when ex vivo expanded cord blood cells are infused as an off-the-shelf non-human leukocyte antigen (HLA) matched product with the goal of providing rapid but transient myelopoiesis in the setting of a single or double umbilical cord blood transplant.

II. Examine the in vivo persistence of the ex vivo expanded cord blood product. The kinetics and durability of hematopoietic reconstitution will be determined and the relative contribution to engraftment of the expanded cord blood product and the unmanipulated cord blood unit(s) in early and long-term engraftment will be determined by frequent determination of donor chimerisms in the peripheral blood.

SECONDARY OBJECTIVES

I. Estimate the incidence and severity of acute and chronic graft-versus-host-disease (GVHD) in patients receiving off-the-shelf ex vivo expanded and cryopreserved cord blood cells.

II. Estimate the incidence of transplant related mortality at day 100.

III. Estimate the incidence of malignant relapse and probabilities of overall and event-free survival at 1 and 2 years post transplant.

IV. Obtain preliminary data on the incidence of infections/viral reactivation from the start of conditioning to 100 days post transplant and then at 6 months, 1 year and 2 years post transplant as possible.

V. Obtain preliminary data on the phenotype and function of immune cells recovering in patients receiving expanded and unmanipulated cord blood grafts.

VI. Examination of possible immunologic factors leading to emergence of a dominant unit.

OUTLINE:

MYELOABLATIVE CONDITIONING: Patients receive fludarabine phosphate intravenously (IV) over 1 hour on days -8 to -6 and cyclophosphamide IV on days -7 and -6. Patients undergo total-body irradiation (TBI) twice daily on days -4 to -1.

TRANSPLANTATION: Patients undergo unmanipulated single- or double-unit umbilical cord blood transplantation on day 0 and receive ex vivo-expanded cord blood progenitor cells IV over 4 hours following the last unmanipulated cord blood infusion.

GVHD PROPHYLAXIS: Patients initially receive cyclosporine (CSP) IV over 1 hour beginning on day -3. CSP may be given orally (PO) when the patient can tolerate oral medications and has a normal gastrointestinal transit time. CSP is given until day 100, and may taper on day 101 if there is no graft versus host disease. Patients also receive mycophenolate mofetil (MMF) IV every 8 hours on days 0 to 7 and then may receive MMF PO beginning day 8 to 30. MMF is continued for a minimum of 30 days or until 7 days after blood counts recover whichever is later. If there is no evidence of acute GVHD and donor cluster of differentiation (CD)3 engraftment is at least 50% from one donor MMF may be tapered.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia:

  * High risk complete response (CR)1 as evidenced by preceding myelodysplastic syndromes (MDS), high risk cytogenetics (for example, monosomy 5 or 7, or as defined by referring institution treatment protocol), >= 2 cycles to obtain CR, erythroblastic or megakaryocytic leukemia; >= CR2
  * All patients must be in CR as defined by hematologic recovery and < 5% blasts by morphology within the bone marrow and a cellularity of >= 15%
  * Patients in which adequate marrow/biopsy specimens cannot be obtained to determine remission status by morphologic assessment, but have fulfilled criteria of remission by flow cytometry, recovery of peripheral blood counts with no circulating blasts, and/or normal cytogenetics (if applicable) may still be eligible; reasonable attempts must be made to obtain an adequate specimen for morphologic assessment, including possible repeat procedures; these patients must be discussed with the Principal Investigator, Colleen Delaney prior to enrollment
* Acute lymphoblastic leukemia:

  * High risk CR1 [for example, but not limited to: t(9;22), t(1;19), t(4;11) or other mixed lineage leukemia (MLL) rearrangements, hypodiploid]
  * Greater than 1 cycle to obtain CR
  * >= CR2
  * All patients must be in CR as defined by hematologic recovery and < 5% blasts by morphology within the bone marrow and a cellularity of >= 15%
  * Patients in which adequate marrow/biopsy specimens cannot be obtained to determine remission status by morphologic assessment, but have fulfilled criteria of remission by flow cytometry, recovery of peripheral blood counts with no circulating blasts, and/or normal cytogenetics (if applicable) may still be eligible; reasonable attempts must be made to obtain an adequate specimen for morphologic assessment, including possible repeat procedures; these patients must be discussed with the Principal Investigator, Colleen Delaney prior to enrollment
* Chronic myelogenous leukemia excluding refractory blast crisis; to be eligible in first chronic phase (CP1) patient must have failed or be intolerant to imatinib mesylate
* Myelodysplasia (MDS) International Prognostic Scoring System (IPSS) intermediate 2 (Int-2) or high risk (i.e., refractory anemia with excess myeloblasts [RAEB], refractory anemia with excess blasts in transformation [RAEB-T]) or refractory anemia with severe pancytopenia or high risk cytogenetics; blasts must be < 10% by a representative bone marrow aspirate morphology
* Karnofsky (>= 16 years old) >= 70%
* Lansky (< 16 years old) >= 50%
* Calculated creatinine clearance must be > 60 mL and serum creatinine =< 2 mg/dL (adults)
* Calculated creatinine clearance must be > 60 mL/min (children < 18 years old)
* Total serum bilirubin must be < 3 mg/dl
* Transaminases must be < 3 x the upper limit of normal
* Diffusion capacity of the lung for carbon monoxide (DLCO) corrected > 50% normal
* For pediatric patients unable to perform pulmonary function tests, oxygen (O2) saturation > 92% on room air
* Left ventricular ejection fraction > 45% OR shortening fraction > 26%
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Uncontrolled viral or bacterial infection at the time of study enrollment
* Active or recent (prior 6 month) invasive fungal infection without infectious disease (ID) consult and approval
* History of human immunodeficiency virus (HIV) infection
* Pregnant or breastfeeding
* If =< 18 years old, prior myeloablative transplant within the last 6 months
* If > 18 years old prior myeloablative allotransplant or autologous transplant
* Extensive prior therapy including > 12 months alkylator therapy or > 6 months alkylator therapy with extensive radiation

Ages: 6 Months to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2010-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Time to neutrophil engraftment | By day 42
  Defined as the first of 2 consecutive days in which the absolute neutrophil count (ANC) >= 500.
Time to platelet engraftment | By day 100
Overall survival | Day 100
Overall survival | Day 180
Overall survival | 1 year
Overall survival | 2 years
Event-free survival | Day 100
Event-free survival | Day 180
Event-free survival | 1 year
Event-free survival | 2 years
Incidence of severe (grades 3-4) acute GVHD | Up to day 100
Incidence of grade greater than or equal to 3 infusional toxicity | By day 100
  Toxicities will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0.
Primary graft failure | By day 42
  Defined as failure to achieve ANC >= 500/mm^3 of donor origin.
Secondary graft failure | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Delaney, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Milano F, Thur LA, Blake J, Delaney C. Infusion of Non-HLA-Matched Off-the-Shelf Ex Vivo Expanded Cord Blood Progenitors in Patients Undergoing Cord Blood Transplantation: Result of a Phase II Clinical Trial. Front Cell Dev Biol. 2022 Apr 4;10:835793. doi: 10.3389/fcell.2022.835793. eCollection 2022. PMID 35445027